CLINICAL TRIAL: NCT06643546
Title: The Effect of Different Simulation Applications Used in Breastfeeding Education on Breastfeeding Knowledge, Skills and Clinical Self-Efficacy of Nursing Students: A Randomized Controlled Trial
Brief Title: Effects of Simulation Practices on Breastfeeding Knowledge and Skills of Nursing Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Sinem Ceylan, RN, PhD, Assistant Prof., Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/95
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Use of Different Simulation Techniques in Breastfeeding Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Experimental): received only theoretical breastfeeding training
  Interventions: Other: theoretical training
- 1st intervention group (Experimental): theoretical breastfeeding training and model simulation training accompanied by scenarios
  Interventions: Other: model simulation training
- 2nd intervention group (Experimental): theoretical breastfeeding training and live simulation training with scenarios
  Interventions: Other: live-simulation

INTERVENTIONS:
Other: theoretical training — received only theoretical breastfeeding training
  Arms: control
Other: model simulation training — theoretical breastfeeding training and model simulation training accompanied by scenarios
  Arms: 1st intervention group
Other: live-simulation — theoretical breastfeeding training and live simulation training with scenarios
  Arms: 2nd intervention group

SUMMARY:
Objective: This study evaluated the effectiveness of breastfeeding education using different simulation techniques on nursing students' breastfeeding knowledge, counseling skills, and clinical self-efficacy.

Method: The study sample consisted of 157 nursing students. Data were collected using a sociodemographic questionnaire, the Breastfeeding Assistance Clinical Preparedness Scale, the Breastfeeding Knowledge Form, the Clinical Self-Efficacy in Performance Scale, and the Breastfeeding Counseling Skills Checklist.

Conclusion: We expect that simulation and standardized patient-based breastfeeding education will effectively improve nursing students' readiness for breastfeeding assistance, breastfeeding knowledge, breastfeeding counseling skills, and clinical self-efficacy in breastfeeding performance.

ELIGIBILITY:
Inclusion Criteria:

having taken a gynecology and obstetrics nursing course, volunteering to participate in the research, and not having received formal training on breastfeeding.

Exclusion Criteria:

voluntarily withdrawing from the research and not participating in any stages of the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Assistance Clinical Readiness Scale | before training, 1 hour after training, 4 weeks after
  In the scale developed by the researchers, students evaluate themselves from 0 (not sure) to 10 (absolutely sure) based on the statement "I am ready to provide breastfeeding counseling and breastfeeding care to a mother who has given birth in the clinic.
Breastfeeding Information Form | before training, 1 hour after training, 4 weeks after
  The Breastfeeding Information Form was prepared by researchers using the breastfeeding information inventory developed by Marzalik in 2004 and the competency verification toolkit guide published by the World Health Organization to ensure the competency of direct care providers in the implementation of the baby-friendly hospital initiative. The form consists of 25 statements. Participants are asked to answer each statement as true, false, and I don't know. A correct answer in the form is worth 1 point, and the highest score on the form is 25 and the lowest is 0. As the score received from the form increases, it is interpreted as the level of breastfeeding knowledge increases. In order to evaluate the appropriateness of the scope and content of the form, expert opinions will be obtained from at least 9 faculty members.
Self-efficacy scale in clinical performance | before training, 1 hour after training, 4 weeks after
  In order to determine the self-efficacy perceptions of nursing students about their clinical performance, the Clinical Performance Self-Efficacy Scale (CPSES) was developed by Cheraghi et al. (2009) in 2009. The Turkish validity and reliability studies of the scale were conducted by Zaybak (2016). The scale, which consists of a total of 37 items, consists of 4 factors (sub-dimensions) as "Data collection", "Diagnosis and planning", "Application" and "Evaluation". The scale's total and sub-dimension score averages are evaluated by taking the item score average. A high score average obtained from the scale indicates that self-efficacy in clinical performance is high. The total Cronbach alpha coefficient of the scale was found to be 0.98.
Breastfeeding Counseling Skills List | 4 week after training
  Created by researchers using professional practice guides. This skill list is used by the student during breastfeeding counseling. Scoring is done based on whether the breastfeeding counseling student demonstrates the skill. There are 25 steps in the skill list. Correct application is evaluated as 2 points, incomplete application as 1 point, and failure to apply as 0 points. The maximum score received from the list is 50 and the minimum score is 0. Expert opinions will be obtained from at least 9 faculty members in order to evaluate the appropriateness of the scope and content of the form

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Nursing Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No